CLINICAL TRIAL: NCT02196948
Title: Electrolysis Percutaneous Therapeutic (EPTE) for the Management of Supraspinatus Tendinopathy
Brief Title: Electrolysis Percutaneous Therapeutic (EPTE) for Supraspinatus Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC 22/2014
Record Dates: First submitted 2014-07-19; First posted 2014-07-22 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Supraspinatus Tendinopathy
Keywords: Supraspinatus, tendinopathy, pain, disability, EPTE
MeSH Terms: conditions — Tendinopathy; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrolysis Percutaneous Therapeutic (EPTE) (Experimental): Electrolysis Percutaneous Therapeutic (EPTE) consists of the application of a galvanic electrical current with an acupuncture needle in the soft tissue, in this case the supraspinatus tendon, to initiate a local inflammatory process allowing phagocytosis and repair of the affected tissue. The technique is pain-free since the electrical intensity is adapted to each patient. In addition, patients will be asked to perform an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles, to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 4 weeks.
  Interventions: Other: Electrolysis Percutaneous Therapeutic (EPTE)
- Eccentric exercise (Experimental): Patients will be asked to perform an eccentric loading exercise program for the shoulder musculature, particularly the supraspinatus and infraspinatus muscles, to be performed on an individual basis twice every day. The therapeutic protocol will be applied for 4 weeks.
  Interventions: Other: Eccentric exercise

INTERVENTIONS:
Other: Electrolysis Percutaneous Therapeutic (EPTE)
  Arms: Electrolysis Percutaneous Therapeutic (EPTE)
Other: Eccentric exercise
  Arms: Eccentric exercise

SUMMARY:
Therapeutic management of supraspinatus tendinopathy is conflicting. There is evidence that eccentric exercise protocols can be effective for this condition. The inclusion of other therapeutic modalities could help to the management of these patients. A new therapeutic approach, called Electrolysis Percutaneous Therapeutic (EPTE) has been clinically developed. The objective of this randomized clinical trial is to determine the effectiveness of the inclusion of EPTE into a eccentric exercise protocol for the management of patients with unilateral supraspinatus tendinopathy

ELIGIBILITY:
Inclusion Criteria:

* Unilateral supraspinatus tendinopathy
* Shoulder pain from at least 3 months
* Shoulder pain of more than 4 points on a NPRS
* Positive findings of supraspinatus tendinopathy on MRI

Exclusion Criteria:

* bilateral shoulder symptoms
* younger than 18 or older than 65 years
* history of shoulder fractures or dislocation
* cervical radiculopathy
* previous interventions with steroid injections
* fibromyalgia syndrome
* previous history of shoulder or neck surgery
* any type of intervention for the neck-shoulder area during the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity before and after the intervention | Baseline, after 2 weeks of treatment and one week after the last session
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area.

SECONDARY OUTCOMES:
Changes in disability before and after the intervention | Baseline, after 2 weeks of treatment and one week after the last session
  The Disabilities of the Arm, Shoulder and Hand (DASH) will be used to determine the disability induced by shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Arias Buría, PT, MSc, Principal Investigator — Hospital Universitario Gregorio Marañón-Universidad Rey Juan Carlos; César Fernández de las Peñas, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain